CLINICAL TRIAL: NCT00358787
Title: Management of Displaced Supracondylar Fractures of the Humerus Using Lateral Versus Cross K Wires: A Prospective Randomized Clinical Trial
Brief Title: Management of Displaced Supracondylar Fractures of the Humerus Using Lateral vs. Crossed K-wires
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kishore Mulpuri, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H04-70532; W04-0180
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Humeral Fractures
Keywords: Supracondylar fracture; humerus; ulnar nerve injury; Baumann's angle; Supracondylar fracture of the humerus
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Crossed K wire orientation for surgical management of a type III Supracondylar fracture.
  Interventions: Procedure: Crossed K-wiring of supracondylar fracture of the humerus
- 2 (Active Comparator): Lateral K wire orientation for surgical management of a type III Supracondylar fracture.
  Interventions: Procedure: Lateral K-wiring of supracondylar fracture of the humerus

INTERVENTIONS:
Procedure: Crossed K-wiring of supracondylar fracture of the humerus — Closed reduction of the fracture followed by crossed K wire percutaneous pinning.
  Arms: 1
Procedure: Lateral K-wiring of supracondylar fracture of the humerus — Closed reduction of the fracture followed by lateral K wire percutaneous pinning.
  Arms: 2

SUMMARY:
Completely displaced (Type III) supracondylar fractures of the humerus are treated in the operating room and are held together with pins stuck into the bone. There are two ways of inserting the pins: crossed and laterally. The crossed method is often used because it is thought to be more stable, but this method also carries a risk of hitting the ulnar nerve. It is not known which method is more stable. Our hypothesis is that loss of reduction will be equivalent between the two pinning methods.

DETAILED DESCRIPTION:
Children with type III supracondylar fractures of humerus who meet the study inclusion criteria will be invited to participate in the study by the on call orthopaedic surgeon. All patients will be required to provide informed consent. Patients will then be randomized through a random number software package and will commence immediately after confirmation of inclusion into the study. The fracture is reduced and fixed percutaneously either with crossed or lateral K wires, according to which group the subject was randomized to. Post reduction antero-posterior and lateral radiographs of the elbow are done in the operating room. Above elbow cast is applied. Radiographs are taken at follow-up visits to the clinic. The radiographs are measured to determine loss of reduction between immediate post-op films and films taken immediately prior to pin removal.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients scheduled for closed reduction and K wiring of supracondylar fractures of the humerus under general anaesthesia a
* Type-3 Supracondylar fractures of the humerus.
* Aged 3 to 7 years old
* Consent to participate in the study

Exclusion Criteria:

* Open supracondylar fractures of the humerus
* Children with pre-operative ulnar nerve injury
* Supracondylar fractures with compartment syndrome needing fasciotomy
* Supracondylar fractures needing vascular repair
* Refusal to provide informed consent

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2008-07; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Loss of reduction between lateral K wires and crossed K wires in the treatment of supracondylar fractures of the humerus (at pin removal)

SECONDARY OUTCOMES:
Functional outcome (3 years post-op) | 3 years
Rate of iatrogenic ulnar nerve injury

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, MD, Principal Investigator — The University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada